CLINICAL TRIAL: NCT05516017
Title: The Effect of Pinhole Glasses on Vestibular Electrical Stimulation Used in the Treatment of Chronic Unilateral Vestibular Hypofunction: A Randomized Controlled Study
Brief Title: The Effect of Pinhole Glasses on Vestibular Electrical Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Huseyin Gezgin, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Istanbul Unversity, Istanbul
Record Dates: First submitted 2022-08-24; First posted 2022-08-25 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Vertigo, Peripheral
Keywords: vestibular electrical stimulation, pinhole glasses
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Electrical Stimulation and exercises with pinhole glasses (Experimental): For VES, which we will apply in our study, the anode will be placed on the mastoid protrusion on the sick ear and a cathode electrode is placed on the healthy ear.The skin to be treated will be cleaned and dried The electrodes are fixed to the head with the help of an elastic band. VES application per session will be applied for 30 minutes, 2 days a week, for 8 weeks. Patients will be asked to perform a bed exercise program once a day for 20-30 minutes each session, 5 days a week, for 8 weeks, including the above exercises, which they will perform in bed after the first day.These exercises are; fixation of the head and turning the eyes to the right and left, the movement of fixing the eyes and turning the head to the left and right, turning the head and eyes in one direction and focusing, hip flexor and knee extensor strengthening.
  Patients in the experimental group will also wear pinhole glasses while applying VES.
  Interventions: Device: Vestibular Electrical Stimulator and Pinhole Glasses
- VES and exercises without pinhole glasses (Active Comparator): For VES, which we will apply in our study, the anode will be placed on the mastoid protrusion on the sick side and the cathode will be placed on the healthy ear. The skin to be treated will be cleaned and dried. The electrodes are fixed to the head with the help of an elastic band. VES application per session will be applied for 30 minutes, 2 days a week, for 8 weeks.Patients will be asked to perform a bed exercise program once a day for 20-30 minutes each session, 5 days a week, for 8 weeks, including the above exercises, which they will perform in bed after the first day.These exercises are; fixation of the head and turning the eyes to the right and left, the movement of fixing the eyes and turning the head to the left and right, turning the head and eyes in one direction and focusing, hip flexor and knee extensor strengthening.
  Patients in the active comparator will not wear pinhole glasses while VES is applied.
  Interventions: Device: Vestibular Electrical Stimulator

INTERVENTIONS:
Device: Vestibular Electrical Stimulator and Pinhole Glasses — It is applied with a vestibular electrical stimulation device for 20 msec with 2 Hz, 1-4 mA, 1 mA increments. Very high frequencies can cause auditory perceptions such as 0.5 - 20 kHz, should be avoided.
  The pinhole glasses are made of 2 pieces of opaque black plastic material with a total of 113 holes on each side. The opaque black plastic is 1.7 mm thick, 4.5 cm wide, and 5.5 cm long.
  The holes in the opaque black material are arranged horizontally in 11 rows from top to bottom. The diameter of each hole is 1.1 mm, the horizontal distance of the holes from each other is 4.5 mm, and the vertical distance is 3.5 mm.
  Arms: Vestibular Electrical Stimulation and exercises with pinhole glasses
Device: Vestibular Electrical Stimulator — It is applied with a vestibular electrical stimulation device for 20 msec with 2 Hz, 1-4 mA, 1 mA increments. Very high frequencies can cause auditory perceptions such as 0.5 - 20 kHz, should be avoided.
  Arms: VES and exercises without pinhole glasses

SUMMARY:
Balance is the ability to control and maintain the body's center of gravity within the support area. One of the important causes of imbalance is right or left sided unilateral vestibular hypofunction. Chronic vestibular hypofunction describes the loss of unilateral peripheral vestibular function lasting more than 3 months. VES is an important method for replacing the sensory afferents lost in the sudden onset of unilateral vestibular hypofunction and for the correct processing of information in the balance center. Regarding the mechanism of action of Vestibular Electrical Stimulation (VES), it is suggested that it generally affects the auditory system at various levels.

Study aimed which was planned as a prospective, randomized, single-blind and single-center study, was conducted between 1 September 2022 and 1 July 2023, to Istanbul University, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Vertigo Rehabilitation Outpatient Clinic with chronic vestibular hypofunction and the inclusion criteria. It was planned to include at least 100 matching patients. Participants who meet the inclusion criteria will be randomized into two groups by computer program after they are numbered according to the order of application. VES and exercise therapy will be applied by wearing pinhole glasses to 50 participants selected to Group 1 (G1-Experimental group). VES and exercise therapy without wearing pinhole glasses in 50 participants selected in Group 2 (G2-Control group) will be applied. Before and after the treatment, the severity of dizziness due to vestibular hypofunction, their emotional state, functionality and physical state and balance status will be evaluated. Dizziness severity will be evaluated with a visual analog scale, and emotional status, functionality and physical condition will be evaluated with the Dizziness Disability Inventory (DHI). Balance status will be determined by Tandem Gait Test, Timed Up and Go Test and Berg Balance Test. Evaluations will be made before treatment, at 1 month of treatment, and at 3 months of treatment (1 month after the end of treatment) by another study blind to treatment.

With the data provided as a result of the research, it has contributed to both our country and the world literature, besides vestibular electrical stimulation, which can be used in the treatment of vestibular hypofunction, we will draw attention to the effectiveness of the use of pinhole glasses.

DETAILED DESCRIPTION:
Balance is the ability to control and maintain the body's center of gravity within the support area. It can be described as a person's ability to stand without falling, even in the most extraordinary situations, and to feel 'good' in his position in space. from the vestibular system, the visual system, and sensory inputs from tactile-propioceptive sources form the organization of our sense of balance. On the other hand, with the participation of the body muscles, motor coordination occurs and in this way, dynamic balance control is provided as well as the completion of afferent inputs. Balance is an active system that works spontaneously and maintaining the posture is one of its biggest goals. Posture in humans is under a complex and intense regulation by the neuromuscular system. Thanks to this regulation, a rapid postural adaptation takes place against changes in the center of gravity during rest and activity. Postural responses that provide this harmony occur with the integration of vestibular, proprioceptive and visual data in the central nervous system. Any disorder in sensory organization and/or motor coordination provided for balance results in 'balance disorder (imbalance)'. One of the important causes of imbalance is right or left sided unilateral vestibular hypofunction. Vestibular hypofunction may be caused by pathologies originating from the vestibular organ located in the petrous part of the temporal bone and/or the vestibular nerve, which carries sensory information from the vestibular organ to the central nervous system. In these pathologies, which can generally be symptomatic from the time of onset, symptoms are often; vertigo, drowsiness, nausea (sometimes with vomiting), postural dysfunction and imbalance. Unilateral vestibular hypofunction; From Ménière's disease, infections with viral agents such as vestibular neuritis or labyrinthitis, vascular etiologies, toxic reactions due to drugs, weakened function of the inner ear due to aging, head trauma that disrupts inner ear structures, brain tumors (acoustic neuroma, etc.) however, it may be caused by surgical interventions or idiopathic processes that do not cause significant structural changes. In patients with acute vestibular loss, severe dizziness, blurred vision, and nausea and vomiting may accompany. Some of the aforementioned causes (such as vestibular neuritis, vestibular labyrinthitis) usually heal after the acute phase without becoming chronic. Chronic vestibular hypofunction describes the loss of unilateral peripheral vestibular function lasting more than 3 months. In these patients, there is a deterioration in image clarity due to balance disorder and rapid head movements, especially on unstable floors or in conditions where visual information is insufficient, which occurs or increases with movement. Vestibular disorders are usually well treated with medical, surgical, or rehabilitative methods. Compensatory mechanisms play an extremely important role in its recovery. The first mechanism in recovery is internuclear inhibition, causing bilateral reduction in vestibular responses, this inhibition should be prevented. The most successful results are obtained with sensory replacement therapy. The main goals of rehabilitation in vestibular hypofunction are; Reducing the failure of the gravitational muscles on the affected side, reducing oscillopsia due to nystagmus, activating the sensory substitution phenomenon, reducing internuclear inhibition, re-activating coordination, reducing spatial disorientation. Exercises applied in vertigo rehabilitation programs; gaze stabilization exercises (adaptation + replacement exercises), postural stability exercises, habituation exercises, relaxation, flexibility, strengthening and proprioception exercises, conditioning exercises. Appropriate exercise is selected depending on the type of vestibular loss, symptoms, and functional capacity. Vestibular Electrical Stimulation Vestibular Electrical Stimulation (VES) with Transcutaneous Electrical Nerve Stimulation (TENS) is the first step in the rehabilitative treatment of acute vertigo.Direct stimulation of vestibular receptors is highly invasive and not suitable in this case, so electrical stimulation of the paravertebral muscles known as vestibular electrical stimulation (VES) is used. Electrical stimulation is a noninvasive method used for the treatment and rehabilitation of unilateral vestibular pathologies in which muscles and nerves are stimulated with surface electrodes. Nerve and muscle stimulation is provided by means of superficial electrodes. Stimulation of peripheral motor nerves and muscles at the same time with TENS can be done by applying electric current to the skin. These are compatible with motor spots. At the same time, the sensory nerves in the skin are also stimulated. This type of stimulation depolarizes the motor nerves either centrifugally or centripedally. Thus, the motor and sensory effects of TENS are seen together. For this reason, it is also used for pain relief. Electrical stimulation with TENS is called Galvanic Electrical Stimulation (GVS), since both are low-frequency currents, although not using galvanic current. GVS is one of the few methods to artificially stimulate the vestibular system. It is mostly applied on the mastoid body, the reason for choosing the mastoid body is because of its proximity to the vestibule in the inner ear. Other artificial methods are caloric and magnetic vestibular stimulation. Since GVS is a more practical and noninvasive method, it is one of the most commonly used types of VES. GVS is a new and highly effective neurorehabilitation method used in many movement disorders. VES is an important method for replacing the sensory afferents lost in the sudden onset of unilateral vestibular hypofunction and for the correct processing of information in the balance center. Regarding the mechanism of action of VES, it is suggested that it generally affects the auditory system at various levels. There is an electrophonic activation of the basilar membrane. There are direct changes in hairy cell receptor potentials. Together, there is a modulation in the transmitter oscillation. It causes changes in the spontaneous activity of the auditory nerve. Modifies cardiovascular autonomic responses. Increases visual spatial abilities. Cognitive function and vestibulospinal reflexes also improve. Auditory illusions present with VES are also affected. It has been shown to suppress tinnitus in some patients. Decreased tinnitus is associated with decreased spontaneous activity in the auditory nerve. All this occurs as a result of the change in cochlear hemostasis. As a result of VES, inner ear reflexes are activated. The use of pinhole glasses, which have an effect on visual field stability by increasing the patient's depth of vision and fixation ability, may increase the effectiveness during VES. However, no study with a similar design was found in the literature review on this subject. Study aimed it was hypothesized that the use of pinhole glasses providing visual focusing, which will be applied in addition to VES, will increase the effectiveness of VES and be effective on vestibular symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral vestibular hypofunction
* Those who complain of dizziness for more than three months
* Meniere's disease
* Age-related vestibular hypofunction
* Sequelae of vestibular neuritis
* Patients diagnosed with vertigo after surgical trauma

Exclusion Criteria:

* Central cause of vertigo (necessary during the examination Neurology and ENT To be evaluated by the department)
* History of orthostatic hypotension, psychosomatic disorder, heart disease, cerebrovascular disease, migraine, tumoral disease
* Advanced cervical spondylosis on direct radiographs (excluded from the outpatient clinic) the future)
* History of major surgical intervention in the head and neck region
* Detection of anemia in complete blood count
* Having more than 6 degrees of myopia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) | Evaluation will be done at baseline (before treatment), at the 1st month and at the 3rd month of the treatment
  It is a scale that shows the degree of impact on quality of life, emotional status and functionality in patients with dizziness and balance disorders. The form developed by Newman and Jacobson includes 25 items that evaluate the problems related to dizziness: 9 questions question functionality, 9 questions emotional state, and 7 questions physical state. Questions are answered by ticking one of the options no, sometimes yes. No answer counts as 0 points, sometimes 2 points and yes answers as 4 points.
Change in Dizziness Severity Evaluated by Visual Analog Scale | Evaluation will be done at baseline (before treatment), at the 1st month and at the 3rd month of the treatment
  It is a subjective measurement made to determine the severity of the patient's dizziness by the patient. For the measurement, the definition of the parameter to be evaluated - the severity of dizziness in our study - is written on the ends of the 10 cm long line and the patients are asked to mark their own condition.

SECONDARY OUTCOMES:
Change in Berg Balance Scale | Evaluation will be done at baseline (before treatment), at the 1st month and at the 3rd month of the treatment
  It is a scale created mainly for the evaluation of balance and determining the risk of falling in the elderly. It consists of 14 items scored between 0-4. The highest possible score is 56. A low score indicates greater risk of falling and loss of balance.
Change in Timed Up and Go Test (TUG) | Evaluation will be done at baseline (before treatment), at the 1st month and at the 3rd month of the treatment
  The patient sits in a chair and a target is set 3 meters ahead. The patient is asked to get up from the chair, walk to the target, come back and sit on the chair again. The elapsed time is recorded. If it lasts longer than 12 seconds, the patient has a risk of falling.
Change in Tandem Walking | Evaluation will be done at baseline (before treatment), at the 1st month and at the 3rd month of the treatment
  The patient is asked to walk on a straight line drawn on the ground, with the toe of one foot touching the heel of the other foot. How many steps he can take is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Karan, Prof Dr., Study Director — Istanbul University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karan A, Alptekin HK, Capan N, Diracoglu D, Saral I, Aydin S, Aksoy C. The efficacy of vestibular electrical stimulation on patients with unilateral vestibular pathologies. Turk J Phys Med Rehabil. 2017 Jun 3;63(2):149-154. doi: 10.5606/tftrd.2017.267. eCollection 2017 Jun. PMID 31453443
- [Result] Rizzo-Sierra CV, Gonzalez-Castano A, Leon-Sarmiento FE. Galvanic vestibular stimulation: a novel modulatory countermeasure for vestibular-associated movement disorders. Arq Neuropsiquiatr. 2014 Jan;72(1):72-7. doi: 10.1590/0004-282X20130182. PMID 24637984